CLINICAL TRIAL: NCT06258005
Title: PocDoc Lipids Study for Increasing Out-of-Surgery Lipid Testing
Brief Title: PocDoc Lipids Out-of-Surgery Study
Status: Completed | Type: Observational
Sponsor: Vital Signs Solutions Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 325988
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PocDoc testing of primary care patients: There are significant numbers of patients in primary care who should be given annual lipid checks who are not receiving them. PocDoc is a digital rapid 5-marker lipid panel that uses a smartphone as a diagnostic reader. PocDoc tests will be offered to patients overdue their annual lipid check either in surgery, in the community or in their own home.
  Interventions: Diagnostic Test: PocDoc
- Pocdoc testing in the community: Providing lipid testing in community settings such as in pharmacy may offer a more attractive solution to consumers. This hypothesis will be tested by offering PocDoc lipid tests in a community setting.
  Interventions: Diagnostic Test: PocDoc
- PocDoc testing in workplaces: Providing lipid testing as part of a health wellness screen in employees workplaces in may offer an attractive solution to consumers needing their lipid levels check. This hypothesis will be tested by offering PocDoc lipid tests as part of corporate wellness screens.
  Interventions: Diagnostic Test: PocDoc

INTERVENTIONS:
Diagnostic Test: PocDoc — PocDoc is a digital rapid 5-marker lipid test

SUMMARY:
This study seeks to improve access to lipid testing in out-of-surgery locations using PocDoc, a UKCA approved IVD device that measures a full 5 marker lipid panel using a smartphone or tablet. The study will investigate whether PocDoc can close the gap in people not tested by exploring 3 new out-of-surgery methods:

1. Lipid testing for high-risk individuals on existing CVD register who have not attended in-surgery appointments
2. Footfall lipid testing conducted in pharmacy or at community events
3. Corporate wellness lipid testing performed by employers for employees as part of an organised corporate wellness check

DETAILED DESCRIPTION:
Lipid testing in out-of-surgery (OOS) locations using a digital lipid measuring device called PocDoc promises to increase access to lipid testing and cardiovascular disease health assessment. PocDoc lipids comprises a smartphone-compatible disposable microchip test strip which uses proprietary colorimetric microfluidic technology to accurately detect lipid biomarkers from a droplet of blood. PocDoc Lipids Professional was launched in 2022 to enable professional users to perform lipid screens as part of lifestyle or preventative healthcare screens. The investigator's hypothesise that providing easier, more cost-effective access to lipid testing at scale, without patients having to attend the GP surgery could:

1. Identify previously unidentified patients (including key "hard to reach" cohorts) who have elevated lipid levels and get them into a lipid lowering clinical pathway which reduces risk of CVD event
2. Enable increase in "treat to target" and move more patients from low / medium intensity statin onto high intensity, which reduces risk of CVD events
3. Identify more cases of undiagnosed FH and getting those patients into a lipid lowering pathway

The SBRI 21 Phase 3 program is funding this collaborative project in partnership with SMASH PCN and AHSN NENC with the objective of increasing access to lipid testing in those geographies.

ELIGIBILITY:
Inclusion Criteria:

* Consent indicated from within PocDoc app
* Subjects are legally competent and capable to understand character, meaning and consequences of the study
* Subjects own an approved mobile device (these will be available at the time of the study on the PocDoc website and the central team will verify individuals have appropriate mobile devices before PocDoc tests are sent to them)

Exclusion Criteria:

* Being unable to give informed consent
* < 18 years or > 85 years
* Legally incompetent
* Language barriers potentially compromising an adequate compliance with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals in the primary prevention setting who have not previously had a cardiovascular event such as a heart attack or stroke as well as individuals in the secondary prevention setting who have had previous cardiovascular events.
Sampling Method: Non-Probability Sample
Enrollment: 4256 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Day 1 - one single test done at one timepoint
  Number and proportion of individuals contacted who conduct a PocDoc test
Achieved response rate | Day 1 - one single test done at one timepoint
  Number and proportion of individuals who conduct a PocDoc test that have dyslipidaemia

SECONDARY OUTCOMES:
PocDoc experience | Day 1 - one single test done at one timepoint
  Number (N) and proportion (%) of individuals reporting a positive experience with the PocDoc testing pathway
PocDoc value | Day 1 - one single test done at one timepoint
  c. Number (N) and proportion (%) of individuals reporting improvements vs in surgery testing procedure with regards to convenience, speed of testing, testing process

CONTACTS AND LOCATIONS:
Locations (1):
- PocDoc Ltd, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No